CLINICAL TRIAL: NCT02055092
Title: A Nordic Multicentre Observational Study of Persons With Young Onset Dementia and Their Families - Factors Influencing Quality of Life, Theirs Specific Needs and the Use of Healthcare Resources
Brief Title: Young Onset Dementia - the Difficult Diagnosis and the Stressful Life for the Whole Family
Status: Completed | Type: Observational
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: The Research Council of Norway (Other); The Hospital of Vestfold (Other); Oslo University Hospital (Other); Sykehuset Innlandet HF (Other); Haraldsplass Deaconess Hospital (Other); Karolinska University Hospital (Other); Copenhagen University Hospital, Denmark (Other); Zealand University Hospital (Other); Landspitali University Hospital (Other); Sykehuset Telemark (Other Government)
Responsible Party: Sponsor
Other Study IDs: 229002
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Frontotemporal Dementia; Alzheimer Disease
Keywords: Young onset dementia; Quality of life; Specific needs; Healthcare resources in dementia; Frontotemporal dementia; Alzheimer's disease; Healthcare services
MeSH Terms: conditions — Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bio samples are collected for analysis and storage in a bio bank as part of the routines for the National Registry of Dementia:
  * Blood plasma and serum for the later analysis of inflammation markers.
  * Whole blood for analysis of apolipoprotein E4-genotype.
  * Cerebrospinal fluid for dementia markers (tau-protein, amyloid).
  * Saliva cortisol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- YOD-FTD: Young onset dementia - frontotemporal dementia, 38 persons with their respective family members.
- YOD-AD: Young onset dementia - Alzheimer's disease, 50 persons with their respective family members.
- LOD: Late onset dementia >= 70 years of age; Control group of 100 persons with dementia (mostly AD and AD/vascular) and their respective family members. Data already collected in a previous study.

SUMMARY:
People diagnosed with young onset dementia are today mostly assigned to the same healthcare services as people developing dementia at an older age. They and their families are however in a quite different life situation, which is likely to generate different challenges and specific needs for tailored healthcare services, of importance in maintaining their perceived quality of life.

The investigators of this study wish to assess the factors influencing these families' quality of life, their specific needs and their use of healthcare services by the use a combination of quantitative and qualitative methods. The main aim of this study is to provide better future healthcare services to these families, and to develop a programme for optimal collaboration between specialist healthcare services and the local dementia teams.

DETAILED DESCRIPTION:
Background: Most common dementia cases in Young Onset dementia (YOD) are Alzheimer's disease (AD) and frontotemporal dementia (FTD). There is little knowledge about the impact on the affected families, especially with regard to FTD. Although their life situation and specific needs differ from that of older people, they are referred to the same healthcare services.

Hypothesis:

1. QoL is poorer among persons with FTD and their families compared to AD at baseline.
2. There is less worsening of QoL after two years in persons with AD and their families compared to FTD.
3. People with YOD have different needs for health care services than older people with dementia.
4. YOD and their families have more unmet needs than older people with dementia.

Methods: Nordic multicenter observational cohort study of YOD-AD and YOD-FTD. 75 persons in each group, living at home with their families, recruited from five Norwegian and four Nordic memory clinics. The control group consists of 100 older people with dementia age ≥70 years. The investigators use a combination of quantitative and qualitative methods.

The follow-up period of the persons with YOD and their family members is two years. Assessments are made at baseline, 12 and 24 months, with telephone check-ups at 6 and 18 months. The main assessment questionnaires are Quality of life in Alzheimer's disease (QoL-AD), Camberwell Assessment of Need in the Elderly (CANE), and Resource Utilization in Dementia Lite (RUD Lite).

Study aims for the quantitative part of the study:

1. To evaluate the quality of life of persons with YOD and their family members.
2. To identify and explore the specific needs of YOD and their families.
3. To assess the use of health resources and calculate the costs associated with care for YOD, in comparison with older persons with dementia.
4. To compare the functional characteristics of YOD with older people with dementia in terms of cognitive decline, impairment of activities of daily living, changes in behavior, and quality of life.

Study aims and methods for the qualitative part of the study:

1. To investigate how people living alone with young-onset dementia cope with everyday life and decision-making. A longitudinal study with qualitative interviews at 6, 12, 24, 36 and 48 months after initial diagnosis
2. To investigate how it is to be a spouse/cohabitation to a person with young-onset of frontotemporal dementia. A retrospective and prospective study with qualitative interviews.
3. To investigate adult children's experiences with the support they received after their parent with young-onset dementia received a dementia diagnose. A retrospective and prospective study with qualitative interviews.
4. To investigate carers of people with young-onset dementia experiences with the support contact service. A longitudinell study study with qualitative interviews.

Results: Inclusion starts Feb 2014. The objective of this study is to ensure optimally tailored service provision and future healthcare planning according to the specific needs of families of YOD, and develop a care programme in collaboration between primary and specialist healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* Debut of dementia symptoms before the age of 65 years, but age at time of inclusion may be up to 70 years.
* FTD (Neary et al 1998 criteria)
* Primary progressive aphasia (Mesulam 2003 criteria)
* AD (DSM-IV)
* Community living, excl. dementia-specific living facilities manned 24/7
* Family member with regular contact at least x 1/week.

Exclusion Criteria:

* Lack of informed consent
* No close or appropriate family member
* Frontal lobe dysfunction due to non-progressive injury, i.e. cerebral infarction
* Frontal lobe dysfunction due to motor neuron disease (ALS)
* Other dementia specific condition with frontal lobe dysfunction (Huntington, HIV, Down syndrome, alcoholic dementia)
* Mental retardation
* Current substance abuse, incl. excessive alcohol consumption for the past 12 months

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: YOD participants are community residing persons recruited from memory clinics in Norway and Nordic countries (Iceland, Sweden and Denmark).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-02; Primary Completion 2017-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Quality of life | Baseline
  Assessments by Quality of Life - Alzheimer's dementia (QoL-AD) and Euroqol-5D (EQ-5D), index person and family member; also by proxy (QoL-AD).
Change from baseline in quality of life at 12 months | Baseline, 12 months
  Assessments by Quality of Life - Alzheimer's dementia (QoL-AD) and Euroqol-5D (EQ-5D), index person and family member; also by proxy (QoL-AD).
Change from baseline in quality of life at 24 months | Baseline, 24 months
  Assessments by Quality of Life - Alzheimer's dementia (QoL-AD) and Euroqol-5D (EQ-5D), index person and family member; also by proxy (QoL-AD).

SECONDARY OUTCOMES:
Specific needs | Baseline
  Assessments by Camberwell Assessment of Need in the Elderly (CANE); 24 items for index person and 2 items for family member needs.
Use of healthcare resources | Baseline
  Assessments by Resource utilization in dementia Lite (RUD Lite).
Cognition | Baseline
  Assessments standardized by the National Registry of Dementia: Mini Mental Status-Norwegian revision (MMSE-NR), Clock drawing Test, Trail making test part A and B, 10-word list memory recall and recognition test, The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) visuospatial figure copying, FAS, Boston Naming Test, Informant questionnaire-on Cognitive decline in Dementia (IQ-CODE).
Neuropsychiatric symptoms | Baseline
  Assessments by Neuropsychiatric Inventory- Questionnaire (NPI-Q).
Activities of Daily Living (ADL) | Baseline
  Assessments by Lawton & Brody I-ADL and Physical Self-maintenance Scale (PSMS).
Relative's stress | Baseline
  Assessments by Relative's Stress Scale (RSS).
Specific needs | 12 months
  Assessments by Camberwell Assessment of Need in the Elderly (CANE); 24 items for index person and 2 items for family member needs.
Specific needs | 24 months
  Assessments by Camberwell Assessment of Need in the Elderly (CANE); 24 items for index person and 2 items for family member needs.
Use of healthcare resources | 12 months
  Assessments by Resource utilization in dementia Lite (RUD Lite).
Use of healthcare resources | 24 months
  Assessments by Resource utilization in dementia Lite (RUD Lite).
Cognition | 12 months
  Assessments standardized by the National Registry of Dementia: Mini Mental Status-Norwegian revision (MMSE-NR), Clock drawing Test, Trail making test part A and B, 10-word list memory recall and recognition test, The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) visuospatial figure copying, FAS, Boston Naming Test, Informant questionnaire-on Cognitive decline in Dementia (IQ-CODE).
Cognition | 24 months
  Assessments standardized by the National Registry of Dementia: Mini Mental Status-Norwegian revision (MMSE-NR), Clock drawing Test, Trail making test part A and B, 10-word list memory recall and recognition test, The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) visuospatial figure copying, FAS, Boston Naming Test, Informant questionnaire-on Cognitive decline in Dementia (IQ-CODE).
Neuropsychiatric symptoms | 12 months
  Assessments by Neuropsychiatric Inventory- Questionnaire (NPI-Q).
Neuropsychiatric symptoms | 24 months
  Assessments by Neuropsychiatric Inventory- Questionnaire (NPI-Q).
Activities of Daily Living (ADL) | 12 months
  Assessments by Lawton & Brody I-ADL and Physical Self-maintenance Scale (PSMS).
Relative's stress | 12 months
  Assessments by Relative's Stress Scale (RSS).
Activities of Daily Living (ADL) | 24 months
  Assessments by Lawton & Brody I-ADL and Physical Self-maintenance Scale (PSMS).
Relative's stress | 24 months
  Assessments by Relative's Stress Scale (RSS).

OTHER OUTCOMES:
Clinical dementia rating | Baseline
  Assessments by Clinical dementia rating scale (CDR) .
Awareness | Baseline
  Assessments by REED scale.
Depressive symptoms | Baseline
  Assessments by Cornell Scale for Depression in Dementia (CSDD) by proxy, and using Geriatric Depression Scale (GDS) and Montgomery-Asberg Depression Rating Scale (MADRS) in family member.
Coping | Baseline
  Assessments by Locus, 17 item, for index person and family member.
Intercurrent disease | 6 months
  Assessments by telephone follow-up interview with index person and family member.
Medication | Baseline
Hospital admission | 6 months
  Assessments by telephone follow-up interview with index person and family member.
Changes in living conditions | 6 months
  Assessments by telephone follow-up interview with index person and family member.
Major life events | 6 months
  Assessments by telephone follow-up interview with index person and family member.
Apo E4-genotype | Baseline
  Whole blood collected at baseline, analysis may be performed at a later stage (stored in research bio bank).
Clinical dementia rating | 12 months
  Assessments by Clinical dementia rating scale (CDR) .
Clinical dementia rating | 24 months
  Assessments by Clinical dementia rating scale (CDR) .
Awareness | 12 months
  Assessments by REED scale.
Awareness | 24 months
  Assessments by REED scale.
Depressive symptoms | 12 months
  Assessments by Cornell Scale for Depression in Dementia (CSDD) by proxy, and using Geriatric Depression Scale (GDS) and Montgomery-Asberg Depression Rating Scale (MADRS) in family member.
Depressive symptoms | 24 months
  Assessments by Cornell Scale for Depression in Dementia (CSDD) by proxy, and using Geriatric Depression Scale (GDS) and Montgomery-Asberg Depression Rating Scale (MADRS) in family member.
Coping | 12 months
  Assessments by Locus, 17 item, for index person and family member.
Coping | 24 months
  Assessments by Locus, 17 item, for index person and family member.
Intercurrent disease | 18 months
  Assessments by telephone follow-up interview with index person and family member.
Medication | 12 months
Medication | 24 months
Medication | 6 months
Medication | 18 months
Hospital admission | 18 months
  Assessments by telephone follow-up interview with index person and family member.
Changes in living conditions | 18 months
  Assessments by telephone follow-up interview with index person and family member.
Major life events | 18 months
  Assessments by telephone follow-up interview with index person and family member.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbæk, MD, PhD, Study Director — Norwegian Centre for Ageing and Health; Hege Kersten, CPh, PhD, Study Chair — Norwegian Centre for Ageing and Health; Aud Johannessen, DrPH, Study Chair — Norwegian Centre for Ageing and Health
Locations (1):
- Norwegian Centre for Ageing and Health, Tønsberg, Vestfold, Norway

REFERENCES:
- [Derived] Hvidsten L, Engedal K, Selbaek G, Wyller TB, Saltyte Benth J, Bruvik F, Kersten H. Quality of life of family carers of persons with young-onset compared to late-onset dementia. Aging Ment Health. 2020 Sep;24(9):1394-1401. doi: 10.1080/13607863.2019.1617245. Epub 2019 May 20. PMID 31106576